CLINICAL TRIAL: NCT00728065
Title: The Effects of Salvia Hispanica-Enriched Foods on Glycemic and Insulinemic Responses and Subjective Satiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Dr. Vladimir Vuksan, Clinical Nutrition and Risk Factor Modification Centre
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 07-121
Record Dates: First submitted 2008-08-01; First posted 2008-08-05 (Estimated); Last update posted 2009-02-18 (Estimated); Status verified 2009-02

CONDITIONS: Post Prandial Blood Glucose

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (10):
- 1 (Experimental): White Bread (control)
  Interventions: Dietary Supplement: White Bread
- 2 (Experimental): White Bread (control)
  Interventions: Dietary Supplement: White Bread
- 3 (Experimental): White bread with 7.32 grams Salba hispanica
  Interventions: Dietary Supplement: White bread with added 7.32g Salvia hispanica
- 4 (Experimental): White bread with 15.58 grams Salba hispanica
  Interventions: Dietary Supplement: White bread with added 15.58g Salvia hispanica
- 5 (Experimental): White bread with 24 grams Salba hispanica
  Interventions: Dietary Supplement: White bread with added Salvia hispanica
- 6 (Experimental): Rice Milk (control)
  Interventions: Dietary Supplement: Rice milk
- 7 (Experimental): Rice Milk (control)
  Interventions: Dietary Supplement: Rice milk
- 8 (Experimental): Rice Milk with 7.32 grams Salba hispanica
  Interventions: Dietary Supplement: Enriched rice milk containing 7.32g Salvia hispanica
- 9 (Experimental): Rice Milk with 15.58 grams Salba hispanica
  Interventions: Dietary Supplement: Enriched rice milk containing 15.58g Salvia hispanica
- 10 (Experimental): Rice Milk with 24 grams Salba hispanica
  Interventions: Dietary Supplement: Enriched rice milk containing 24g Salvia hispanica

INTERVENTIONS:
Dietary Supplement: White Bread — About 100g of white bread consisting of 50g of available carbohydrates, served with 250mL water
  Arms: 1; 2
Dietary Supplement: White bread with added 7.32g Salvia hispanica — About 100g of white bread consisting of 50g of available carbohydrates and 7.32g Salvia hispanica, served with 250mL water
  Arms: 3
Dietary Supplement: White bread with added 15.58g Salvia hispanica — About 100g of white bread consisting of 50g of available carbohydrates and 7.32g Salvia hispanica, served with 250mL water
  Arms: 4
Dietary Supplement: White bread with added Salvia hispanica — About 100g of white bread consisting of 50g of available carbohydrates and 24g Salvia hispanica, served with 250mL water
  Arms: 5
Dietary Supplement: Rice milk — Rice milk containing 50g of available carbohydrates
  Arms: 6; 7
Dietary Supplement: Enriched rice milk containing 7.32g Salvia hispanica — Rice milk containing 50g of available carbohydrates with 7.32g added Salvia hispanica
  Arms: 8
Dietary Supplement: Enriched rice milk containing 15.58g Salvia hispanica — Rice milk containing 50g of available carbohydrates with 15.58g added Salvia hispanica
  Arms: 9
Dietary Supplement: Enriched rice milk containing 24g Salvia hispanica — Rice milk containing 50g of available carbohydrates with 24g added Salvia hispanica
  Arms: 10

SUMMARY:
Salvia hispanic (Salba) is postulated to increase satiety. This study determines the optimal amount of Salba as well as whether liquid or solid enriched products will produce maximum satiety. The results can gauge the effectiveness of Salba in weight loss programs. The study has a randomized, double-blind crossover design which includes 10 test meals and capillary blood sampling to perform glucose and insulin analyses (to determine blood glucose response and blood insulin response).

DETAILED DESCRIPTION:
There are many factors that are involved in the ability of foods to suppress appetite, for instance the fiber, fat and protein contents of the food. The novel whole grain Salvia hispanica may significantly lower appetite compared to refined carbohydrates and other whole grains because of its composition. First, Salvia hispanica's high fiber content may help lower postprandial glycemia. Whole grains are much higher in fiber than refined carbohydrates. High fiber foods are thought to be more satiating because they have lower energy densities and delay gastric emptying, causing glucose to be released more slowly into the circulation. This, in turn, is hypothesized to increase satiety by preventing a sudden drop in blood glucose levels, which would normally trigger hunger . Another mechanism by which fiber may promote satiety, independent of glycemic responses, is through the secretion of gut hormones that signal fullness . Furthermore, Salvia hispanica may be more satiating than other whole grains due to its higher fat and protein contents. Protein and fat also prolong satiety due to mechanisms such as delayed gastric emptying and secretion of gut hormones .

Results from preliminary studies confirm the satiating effects of Salvia hispanica, as they demonstrate that this grain induces increased subjective satiety and reduced postprandial glycemia. It is presumed that if a food is satiating, it will decrease subsequent intake of other foods because hunger is suppressed. A lower caloric intake, in turn, would help promote weight loss.

Salvia hispanica may also encourage weight loss via another mechanism. Preliminary studies suggested that this grain has a lower glycemic index value than white flour. Consumption of low-GI foods compared to high-GI foods has been suggested to reduce obesity by discouraging fat deposition and promoting fat oxidation . Thus, Salvia hispanica could potentially promote weight loss by reducing both hunger and the amount of body fat stored.

In order to study Salvia hispanica's ability to promote weight loss, feasibility studies must first be done to determine what amount is optimal for satiety and also whether enriched products are most satiating in liquid or solid form.

ELIGIBILITY:
Inclusion Criteria:

* BMI 20-35 kg/m2

Exclusion Criteria:

* Endocrine disease (adrenal disorders, glucose homeostasis disorders, metabolic bone diseases, pituitary gland disorders, parathyroid gland disorders, thyroid disorders)
* Pregnancy
* Use of drugs that influence carbohydrate metabolism (e.g. systemic glucocorticoids, beta blockers, thiazide diuretics)
* Use of fiber supplements
* Substance abuse (including regular smoking)
* Digestive or malabsorption disorders (malabsorption syndrome, Crohn's disease, stomach ulcer, duodenal ulcer or intestinal parasites)
* Presence of any significant disease or condition, including emotional or psychiatric disorders, that, in the opinion of the investigator, is likely to alter the metabolic state or interfere with the subject's ability to complete the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2007-12; Primary Completion 2008-09 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Post prandial capillary blood glucose levels | 2 hour period, Every 15 minutes for first hour, every 30 minutes for second hour

SECONDARY OUTCOMES:
Patient completed satiety questionnaire | 2 hour period, Every 15 minutes for first hour, every 30 minutes for second hour

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Nutrition and Risk Factor Modification Centre, Toronto, Ontario, Canada